CLINICAL TRIAL: NCT04032665
Title: Reveal Transition: Rivaroxaban-Evaluation of Variables Enhancing Antithrombotic Efficacy and Longterm-Outcome in Stabilized Patients With Cardiovascular Disease. A Mechanistic Study in Transition / Stabilized Phase of CAD
Brief Title: Reveal Transition - A Mechanistic Study in Transition / Stabilized Phase of CAD
Acronym: RevealTrans
Status: Withdrawn | Type: Observational
Why Stopped: study design reconsidered
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: Reveal Transition
Record Dates: First submitted 2019-07-18; First posted 2019-07-25 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2019-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stable coronary and peripheral artery disease (CAD/PAD): Stable CAD/PAD patients with previous percutaneous coronary intervention and drug eluting stent-implantation treated with dual antiplatelet therapy (ASA+clopidogrel)
  Interventions: Diagnostic Test: Rivaroxaban
- Acute coronary artery disease (ACS): Patients with troponin-positive ACS (NSTEMI/STEMI) with planned percutaneous coronary intervention and drug eluting stent-implantation treated with P2Y12 inhibitor (ticagrelor) and ASA
  Interventions: Diagnostic Test: Rivaroxaban

INTERVENTIONS:
Diagnostic Test: Rivaroxaban — In stable CAD/PAD patients with previous PCI and DES-implantation treated with DAPT (ASA+clopidogrel) platelet rich plasma (PRP) and washed platelets as well as serum/plasma/urinary samples will be collected between 2 and 4 weeks before switching from DAPT to ASA + rivaroxaban (2,5 mg b.i.d.), between 2 and 4 weeks under monotherapy with ASA 100mg o.d., and between 2 and 4 weeks under therapy with ASA 100mg o.d. + rivaroxaban (2,5 mg b.i.d.) and treated ex vivo with rivaroxaban to asses platelet activation and function, platelet-triggered thrombin generation and platelet-dependent vascular inflammation.

SUMMARY:
Longterm oral anticoagulation with very low dose rivaroxaban (2.5mg bid) in combination with aspirin has been shown superior over standard aspirin monotherapy in patients with stable coronary artery disease (CAD) in the COMPASS trial. To date, there are no data comparing these - antithrombotic strategies and to provide insights about mechanistic effects of very low dose rivaroxaban on top of aspirin for longterm treatment.

Thus, the goal of the planned pilot study will be to identify effects of rivaroxaban on platelet function, platelet-mediated vascular inflammation and particularly, platelet-mediated thrombin generation as well as the underlying mechanisms and to reveal differences in mechanistic effects during longterm treatment with combined novel antiplatelet/anticoagulant strategies. This study is planned as descriptive study.

ELIGIBILITY:
Inclusion Criteria:

1. patients≥ 18 years.
2. troponin-positive acute coronary syndrome (NSTEMI/STEMI) with planned dual antiplatelet therapy (DAPT, ASA + ticagrelor) for 12 months or stable CAD with previous PCI and drug eluting-stent (DES) + pre-existing PAD under treatment with DAPT (ASA + clopidogrel).
3. Patients with coronary artery disease who are younger than 65 years of age are required to have documentation of atherosclerosis involving at least two vascular beds or to have at least two additional risk factors (current smoking, diabetes mellitus, an estimated glomerular filtration rate [GFR] <60 ml per minute, heart failure, or nonlacunar ischemic stroke ≥1 month earlier).
4. informed written consent.

Exclusion Criteria:

1. any condition that requires longterm or already ongoing full oral anticoagulation (e.g. recent systemic embolism, prosthetic heart valves or chronic atrial fibrillation).
2. patients with increased bleeding risk preventing guideline adherent dual antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients post troponin-positive acute coronary syndromes (STEMI n=17 + NSTEMI n=17) or stable CAD + peripheral artery disease (PAD) (n=17) with additional risk factors (see inclusion cirteria) who underwent PCI.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Inflammation, Thrombogenicity and Mechanistic Insights During Transition from acute to chronic phase | 2 years
  Define the course of vascular inflammation and thrombogenicity during transition from acute to chronic phase after percutaneous coronary intervention and to provide mechanistic insights of very low dose rivaroxaban (VLDR) on platelet activation and function, platelet-triggered thrombin generation and platelet-dependent vascular inflammation. Platelet function as well as platelet-dependent vascular inflammation will be determined by flow cytometry, thrombinoscopy, spectrofluorimetry, aggregometry, total thromus-formation analysis system (T-TAS) and thrombelastography (TEG) studies

SECONDARY OUTCOMES:
Biomarker Expression | 2 years
  To reveal course of prothrombotic and inflammatory markers after acute coronary syndromes to better understand the transition from acute to stabilized phase.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Geisler, Professor, Principal Investigator — University Hospital of Tuebingen; Oliver Alexander Borst, Professor, Principal Investigator — University Hospital of Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No